CLINICAL TRIAL: NCT02673749
Title: A Phase 2b/3, Multicenter, Randomized, Double-Blind, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy, Safety, and Tolerability of Two Doses of RP-G28 in Subjects With Lactose Intolerance
Brief Title: Efficacy, Safety, and Tolerability Study of RP-G28 in Subjects With Lactose Intolerance
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ritter Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G28-003
Record Dates: First submitted 2016-01-25; First posted 2016-02-04 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2017-04

CONDITIONS: Lactose Intolerance
Keywords: Lactose maldigestion; Dairy intolerance; Intolerance to milk; Intolerance to dairy; Milk intolerance; GI disorder; Lactose metabolism; GI symptoms after dairy ingestion
MeSH Terms: conditions — Lactose Intolerance | interventions — RP-G28

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- RP-G28 Dose 1 (Experimental)
  Interventions: Drug: RP-G28
- RP-G28 Dose 2 (Experimental)
  Interventions: Drug: RP-G28
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: RP-G28 — Study drug taken orally
  Arms: RP-G28 Dose 1; RP-G28 Dose 2
Other: Placebo — Placebo taken orally
  Arms: Placebo

SUMMARY:
RP-G28 is being investigated for treatment of moderate to severe lactose intolerance and its potential to improve the tolerance of lactose (dairy products).

DETAILED DESCRIPTION:
Lactose intolerance is a common gastrointestinal (GI) disorder that develops in lactose maldigesters when consuming lactose or when lactose is added to a previously low-lactose diet. Lactose intolerance is characterized by one or more of the cardinal symptoms that follow the ingestion of lactose-containing foods. These symptoms include; abdominal pain, cramping, bloating, flatulence [gas] and diarrhea. As such, most lactose intolerant individuals avoid the ingestion of milk and dairy products, while others substitute non-lactose containing products in their diet. Currently, there are no approved treatments for this condition.

Based on the health implications from insufficient calcium intake over a lifetime, including increased risk of osteoporosis and hypertension, there is need in the medical community for a tolerable and convenient treatment that allows for all levels of milk and dairy product consumption in people suffering from mild to severe lactose intolerance.

Study Objective:

To access efficacy of two RP-G28 dosing regimes on symptoms related to lactose intolerance relative to placebo after 30 days of treatment. The 30 day post-treatment phase will further evaluate the treatment's potential to prolong relief from symptoms.

Study Design:

The participants will take about 60 days to complete the study. The study consists of 3 distinct phases: Screening, a 30-day Treatment Phase, and a 30-day Post-Treatment Phase (off study treatment observation period). A participant will need to visit the clinical only 6 times throughout the study.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

* Female subjects must be non pregnant, and non lactating. Females of childbearing potential must use adequate birth control during study participation
* Medical history of intolerance to milk and other dairy products, and/or confirmed physician diagnosis of lactose intolerance.
* Must be free from any disorder known to be associated with gastrointestinal disease: irritable bowel syndrome (IBS), inflammatory bowel disease (IBD), ulcerative colitis (UC), Crohn's disease (CD), Celiac disease, diverticulitis, chronic constipation, chronic pancreatitis, pancreatic insufficiency, symptomatic biliary disease, small intestine bacterial overgrowth syndrome (SIBO), active gastric or duodenal ulcers, or history of severe ulcers.
* Must be nicotine free.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2016-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in abdominal pain | Day 31
  Percent change from baseline to Day 31 of AUC abdominal pain symptom score based on measures taken after a lactose challenge test at 1, 2, 3, 4, and 5 hours. The method of assessment for this outcome measure is an 11-point numeric rating scale completed by the subject.

CONTACTS AND LOCATIONS:
Locations (1):
- Covance, Inc., Princeton, New Jersey, United States

REFERENCES:
- [Derived] Azcarate-Peril MA, Roach J, Marsh A, Chey WD, Sandborn WJ, Ritter AJ, Savaiano DA, Klaenhammer TR. A double-blind, 377-subject randomized study identifies Ruminococcus, Coprococcus, Christensenella, and Collinsella as long-term potential key players in the modulation of the gut microbiome of lactose intolerant individuals by galacto-oligosaccharides. Gut Microbes. 2021 Jan-Dec;13(1):1957536. doi: 10.1080/19490976.2021.1957536. PMID 34365905